CLINICAL TRIAL: NCT01316172
Title: A Prospective, Randomized Controlled Study Demonstrating a Novel, Effective Model of Communication Among Physicians: The 5 Cs of Consultation
Brief Title: Consultation in the Emergency Department
Acronym: 5 Cs
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Health Services Research
Other Study IDs: 2009-0499
Record Dates: First submitted 2011-03-15; First posted 2011-03-16 (Estimated); Last update posted 2019-08-08 (Actual); Status verified 2019-08

CONDITIONS: Communication
Keywords: consultation
MeSH Terms: conditions — Communication

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 5 Cs (Experimental): Educational intervention
  Interventions: Behavioral: 5 Cs
- Control (No Intervention)

INTERVENTIONS:
Behavioral: 5 Cs — education on consultation
  Arms: 5 Cs

SUMMARY:
This study intends to evaluate consultation in the Emergency Department. The purpose is to demonstrate that standardizing communication in the Emergency Department may lead to improved consultation.

ELIGIBILITY:
Inclusion Criteria:

* Emergency medicine residents (PGY1-5)

Exclusion Criteria:

* Did not want to partake in the study

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2010-05; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Consultation effectiveness as measured by global rating scale | Up to 2 weeks
  A global rating scale will be used to measure effectiveness of the intervention.

SECONDARY OUTCOMES:
Consultation effectiveness as determined by a Checklist rating | 2 weeks
  The checklist will be based off of the educational intervention, the 5 Cs, and the global rating scale will be based on expert assessment.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Illinois-Chicago, Chicago, Illinois, United States

REFERENCES:
- [Derived] Kessler CS, Afshar Y, Sardar G, Yudkowsky R, Ankel F, Schwartz A. A prospective, randomized, controlled study demonstrating a novel, effective model of transfer of care between physicians: the 5 Cs of consultation. Acad Emerg Med. 2012 Aug;19(8):968-74. doi: 10.1111/j.1553-2712.2012.01412.x. PMID 22905961